CLINICAL TRIAL: NCT03168724
Title: Efficacy Potential of Goal Management Training to Improve Cognitive Function in Older People Living With HIV
Brief Title: Goal Management Training, Executive Functions and HIV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Marie-Josée Brouillette, Associate Professor, McGill University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MUHC-16-031
Record Dates: First submitted 2017-04-28; First posted 2017-05-30 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Hiv
Keywords: Cognition; Intervention; Self-management; Rehabilitation
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GMT Intervention (Experimental): Over the course of 9 weeks, there are 2h-group sessions with a therapist.
  Interventions: Behavioral: GMT intervention
- Control (No Intervention): Group not getting the intervention

INTERVENTIONS:
Behavioral: GMT intervention
  Arms: GMT Intervention

SUMMARY:
Goal Management Training (GMT) is a cognitive rehabilitation program targeting executive dysfunction (problems with attention, reasoning, problem solving, planning, etc), which is a central problem in HIV-associated neurocognitive disorder. It teaches self-management principles, stress management and mindfulness, and trains participants in the use of several strategies to reduce cognitive load in everyday tasks, and methods to cue attention to maintain focus on specific tasks. GMT is a manualized protocol with set content conveyed through a combination of slides and a workbook. Two-hour small group sessions are led, in person, by a trained therapist once a week, for nine weeks. The small group sessions allow participants to learn from each other, enhancing engagement. GMT has been shown to improve cognitive function in a variety of neurological conditions, as well as in healthy older people with cognitive concerns. These improvements have been shown to last at least 6 months in some studies and are accompanied by changes in the brain networks underlying executive function. GMT is thus a well-validated, high yield intervention with which to test the potential of cognitive rehabilitation in older HIV+ people with cognitive concerns.

The researchers hypothesize that GMT will lead to improved cognitive function as assessed by better performance on cognitive tests and reduced self-reported cognitive difficulties in people with stable HIV infection who report cognitive difficulties at baseline.

DETAILED DESCRIPTION:
Rehabilitation is a well-established approach to maintain function in the face of chronic disease, and holds promise for addressing the health challenges faced by older people with HIV. A Canadian-led knowledge synthesis review published in 2014 identified cognitive rehabilitation as a promising approach in HIV, but highlighted the absence of high quality, HIV-specific evidence in this area. A recent focused review also highlights the dearth of evidence on this topic. Very few studies have been published, and to date all have been restricted to computerized training programs only. While there is limited evidence for computerized cognitive rehabilitation in any context, there is better evidence for more conventional, in-person rehabilitation approaches, at least in other neurological disorders. Although computerized training is appealing because it is more feasible to deliver on a wide scale than conventional cognitive rehabilitation, The researchers propose that the first step should be to establish an evidence base regarding the efficacy of any form of cognitive rehabilitation in HIV. Evidence of efficacy of a 'high dose' established rehabilitation method could be followed by work to define the key elements, and to study how those elements could be delivered most cost-effectively, but there is no point in pursuing these secondary steps if the most well-established cognitive rehabilitation approaches do not show efficacy. Thus, the researchers propose to test conventional rehabilitation as a crucial first step is a research program focused on evidence-based interventions for improving brain health in HIV.

There is no gold standard conventional cognitive rehabilitation program, but most existing approaches combine face-to-face therapy with at home practice over a period of at least several weeks. In the absence of a gold standard, the researchers have selected one such program: Goal Management Training (GMT). This program targets executive dysfunction, which is a central problem in HIV-associated neurocognitive disorder. GMT is grounded in a neurobiological framework and was developed based on nearly two decades of research on practical approaches to minimizing the impact of executive dysfunction, aiming to help people with brain injury manage real life tasks. The program teaches self-management principles, stress management and mindfulness, and trains participants in the use of several explicit strategies to reduce cognitive load in everyday tasks, and methods to cue attention to maintain focus on specific tasks. GMT is a manualized protocol with set content conveyed through a combination of slides and a workbook. Two-hour small group sessions are led, in person, by a trained therapist once a week, for seven weeks. The small group sessions allow participants to learn from each other, enhancing engagement. GMT has been shown to improve cognitive function in a variety of neurological conditions, as well as in healthy older people with cognitive concerns. Evidence from randomized trials shows that this intervention leads to (i) significant improvements in performance on cognitive tests, including naturalistic tests of real life tasks, (ii) reduced self-reported cognitive difficulties, and (iii) significant improvements in everyday function compared to either a wait-list condition or a general brain health education control. Positive effects have been found in older people with cognitive difficulties, and neurological populations with mild cognitive impairment including mild traumatic brain injury, stroke and spina bifida. These improvements have been shown to last at least 6 months in some studies and are accompanied by changes in the brain networks underlying executive function. GMT is thus a well-validated, high yield intervention with which to test the potential of cognitive rehabilitation in older HIV+ people with cognitive concerns.

The pilot project is nested within an ongoing observational cohort study that aims to understand and address the heterogeneous, multi-factorial nature of compromised brain health in people living with HIV. Study participants will be randomly selected from those participating in the ongoing, longitudinal Positive Brain Health Now (+BHN) study at 2 sites in Montreal (The Montreal Chest Institute and L'Actuel Medical Clinic). This CIHR Team Grant-supported observational, prospective cohort study has enrolled 840 consecutive patients attending 5 HIV clinics across Canada, who are followed every 9 months for 27 months.

Procedure Participants will be recruited either at the time of their routine +BHN study visit, or by phone or by email. Informed consent will occur with the therapist during the first GMT group session during which they will also complete a questionnaire regarding any cognitive concerns they may have (Communicating Cognitive Concerns-C3Q). At the end of the last GMT session, they will be asked to complete the C3Q again. Then, within 4 weeks of completing the GMT program, they will be asked to repeat the B-CAM, coincident with the +BHN study visit if timing permits.

Intervention The standard GMT program lasts 9 weeks and involves 9 weekly 2-hour small group sessions led by a trained therapist. It follows a manualized program that teaches participants a series of techniques to build attention and executive function, and shows them how to implement these techniques in their everyday life. The small group sessions allow individualization of the training to show how it can be applied to meet the particular challenges reported by participants, and explicitly encourage participants to share their challenges and successes with others in the group to promote learning and engagement with the program. The sessions are reinforced with homework, in which participants practice what they have learned. Sessions will be audiotaped for later review by the trainer and/or study investigators to ensure adherence to the intervention manual. The material, including homework, is provided in a workbook that participants use throughout the training, and keep for later reference.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection for at least 1 year
* Able to communicate in French or English
* Capable of providing informed consent
* Over 45 years old
* Subjective cognitive complaints
* Performance on objective computerized cognitive tests that falss at or below 50th percentile of performance in the cohort (main study) as a whole)

Exclusion Criteria:

* Presence of dementia
* Life expectancy of 3 years or less
* Other neurological disorder including opportunistic CNS infection, psychotic disorder
* Current substance dependence or abuse
* Hepatitis C requiring interferon therapy during the study period

Min Age: 46 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Performance measure (B-CAM) | Up to 9 months before the intervention and up to 2 months after the intervention
  We will be looking at changes on the B-CAM (brief cognitive ability measure) pre- and post-intervention

SECONDARY OUTCOMES:
Tower of London (cognitive outcome measure) | Up to 9 months before the intervention and up to 2 months after the intervention
  Assesses planning and mental flexibility
Communicating Cognitive Concerns (C3Q) | On the first day of the intervention and 9 weeks after the beginning of the intervention
  Evaluates cognitive concerns participants may have

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Josee Brouillette, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Lesley Fellows, MD/PhD, Principal Investigator — McGill University
Locations (2):
- Canada (2):
  - Clinique Medicale L'Actuel, Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-07): https://cdn.clinicaltrials.gov/large-docs/24/NCT03168724/Prot_SAP_000.pdf